CLINICAL TRIAL: NCT05017090
Title: Ultrasound-guided Bilateral Modified-thoracoabdominal Nerves Block Through a Perichondrial Approach in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Analgesic Effect of Ultrasound-guided Bilateral Modified-thoracoabdominal Nerves Block Through a Perichondrial Approach
Acronym: M-TAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-2021/09
Record Dates: First submitted 2021-08-15; First posted 2021-08-23 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-08

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Modified-thoracoabdominal nerves block; Acute pain; laparoscopic cholecystectomy
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator) Blocks will be administered after induction of general Anesthesia so participants will be blinded to which intervention they have had.
  Study investigators will not be aware of what group the participant belongs to when assessing the patient at post-operative period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Sham Comparator): The patients in Group N will not receive any intervention. In the intervention and control groups, block sites will be covered with dressings, and patients and other health care workers will be blinded to treatment allocation. The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, tenoxicam, and tramadol.
  Interventions: Other: Standard perioperative and postoperative multimodal analgesia
- Group M-TAPA (Experimental): After tracheal intubation, a high-frequency linear probe will be placed in the sagittal direction at the 10th costal margin, and transversus abdominis, internal oblique, and external oblique muscles will be identified. A block needle will be inserted with in-plane technique and 25 ml 0.25 bupivacaine will be applied to the lower aspect of the chondrium. The same procedure will be repeated on the contralateral side. The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, tenoxicam, and tramadol.
  Interventions: Procedure: M-TAPA block; Other: Standard perioperative and postoperative multimodal analgesia

INTERVENTIONS:
Procedure: M-TAPA block — After tracheal intubation, a high-frequency linear probe will placed in the sagittal direction at the 10th costal margin, and transversus abdominis, internal oblique, and external oblique muscles will be identified. A block needle will inserted with in-plane technique and 25 ml 0.25 bupivacaine will be applied to the lower aspect of the chondrium. The same procedure will be repeated on the contralateral side.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Followup and Monitorization
  Arms: Group M-TAPA
Other: Standard perioperative and postoperative multimodal analgesia — The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). Patients will receive standard multimodal analgesia comprising paracetamol, tenoxicam, and tramadol.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Followup and Monitorization

SUMMARY:
This study will define the postoperative analgesic effect of ultrasound-guided bilateral modified-thoracoabdominal nerves block through perichondrial approach (M-TAPA) and compare the control group in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the most common laparoscopic procedure and causes moderate to severe postoperative pain. The M-TAPA block was described by Tulgar et al. for postoperative analgesia of abdominal surgeries. However, studies showing the analgesic efficacy of this block are lacking. In this prospective interventional trial, the investigators aim to define the efficacy of M-TAPA block for laparoscopic cholecystectomy surgeries under general anesthesia.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective laparoscopic cholecystectomy will be screened for enrollment in the study. After randomization, the patients in the Group M-TAPA will receive bilateral M-TAPA block at the beginning of the operation defined by Tulgar et al or no intervention (Group N). An anesthesiologist who performed M-TAPA block will not involve in the data collection. Other health care workers who will involve in the evaluation of postoperative pain scores, vital parameters, nausea and vomiting, anti-emetic and opioid consumption will be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age between 18 and 70 years with American Society of Anesthesiology (ASA) physical status I-II, who will be scheduled for an elective laparoscopic cholecystectomy surgery included in the study

Exclusion Criteria:

* presence of coagulation disorder
* refuse to participate
* infection at the injection site of the block
* known allergy to local anesthetics
* advanced hepatic or renal failure
* can not communicate in Turkish
* history of abdominal surgery or trauma
* conversion of laparoscopic to open surgery
* consumption of any pain killers within the 24 h before the operation
* chronic opioid consumption
* pregnancy
* alcohol or drug abuse
* body mass index (BMI) ≥ 35 kg m-2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale scores | 24 hours
  The primary outcome variable is Numerical Rating Scale scores both at rest and motion. A blinded anesthesiologist will assess postoperative pain during rest and motion at the postoperative 15th,30th and 60th minute, second,6th, 12th and 24th hour by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable).

SECONDARY OUTCOMES:
Opioid consumption | 24 hours
  If NRS score of the patient is equal or over 4, IV 50 mg tramadol will be applied as a rescue analgesic.
Adverse events | 24 hours
  Incidence of nausea and vomiting during postoperative 24 hour time period will be noted.
Metoclopromide consumption | 24 hours
  The severity of the nausea will be assessed on a 4 -point scale (0=none 1=mild, 2=moderate 3=severe). If the patients nausea score is ≥2 the patient will receive 10 mg metoclopromide.
Sedation score | 24 hours
  Sedation level of the patients will be assessed on a 4-point scale (0=alert, 1=sleepy, easy to arouse verbally, 2= drowsy, 3=does not open eyes to verbal commands) at postoperative 15th,30th and 60th minute, second,6th, 12th and 24th hour.
Quality of recovery levels between groups by using QoR-40 questionnaire | Postoperative 24th hour
  QoR-40, a 40-item questionnaire that provides a global score and sub-scores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200.Global QoR-40 scores range from 40 to 200 representing, respectively, very poor to outstanding quality of recovery. QoR-40 score will be recorded on the morning of operation and at the postoperative 24th hour.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD, DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)